CLINICAL TRIAL: NCT02086968
Title: Multicenter Randomized Open-label Controlled Study to Investigate Treatment Response of IV Injectafer vs Oral Iron to Baseline Hepcidin Levels in Patients With Iron Deficiency Anemia Secondary to Inflammatory Bowel Disease or Gastric Bypass
Brief Title: Treatment Response of Injectafer vs Oral Iron to Baseline Hepcidin Levels in Patients With Iron Deficiency Anemia (IDA) Secondary to Inflammatory Bowel Disease (IBD) or Gastric Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT13035
Record Dates: First submitted 2014-03-12; First posted 2014-03-13 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Iron Deficiency Anemia Secondary to IBD or Gastric Bypass
MeSH Terms: interventions — ferric carboxymaltose; Iron-Dextran Complex; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Injectafer (Active Comparator): 2 doses of Injectafer, at 15 mg/kg for a maximum single dose of 750 mg given on Days 0 and 7 for a total of up to 1500 mg
  Interventions: Drug: Injectafer
- Ferrous Sulfate tablets (Active Comparator): Oral Ferrous Sulfate at 325 mg (1 tablet) three times a day for 28 days
  Interventions: Drug: Ferrous Sulfate tablets

INTERVENTIONS:
Drug: Injectafer — 2 doses of Injectafer, at 15mg/kg for a maximum single dose of 750mg given on days 0 and 7 for a total of up to 1500mg
  Other Names: Ferric Carboxymaltose (FCM)
  Arms: Injectafer
Drug: Ferrous Sulfate tablets — 325mg (1 tablet) three times a day for 28 days
  Other Names: Oral Iron tablets
  Arms: Ferrous Sulfate tablets

SUMMARY:
The primary objective of this study is to evaluate the treatment response of Injectafer vs. oral iron to baseline hepcidin levels to determine if any of these select IBD or Gastric Bypass patients may demonstrate to be inappropriate for oral iron therapy.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the treatment response of Injectafer vs. oral iron in patients with varying hepcidin levels correlating the treatment response/hepcidin levels to more common laboratory parameters such as ferritin and CRP (C-Reactive Protein) levels and possibly determine if any of these select IBD or Gastric Bypass patients may demonstrate to be inappropriate for oral iron therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female subjects ≥ 18 years of age with clinical diagnosis of IDA secondary to IBD or Gastric Bypass
* Screening Hemoglobin (Hb) ≤ 11g/dL
* Screening Ferritin ≤ 100 ng/mL
* Female subjects who are of childbearing age must have a negative pregnancy test at screening and be practicing an acceptable method of birth control during the study

Exclusion Criteria:

* Hypersensitivity reaction to any component of IV Injectafer or oral iron
* Requires dialysis for treatment of chronic kidney disease (CKD)
* During the 30 day period prior to screening has been treated with IV iron
* No evidence of iron deficiency
* During the 30 day period prior to screening has been treated with a red blood cell transfusion.
* Any non-viral infection
* Known positive hepatitis with evidence of active disease
* Received an investigational drug within 30 days of screening
* Active malignancy within 5 years. Basal or squamous cell skin cancer is not exclusionary
* Alcohol or drug abuse within the past 6 months
* Hemochromatosis or other iron storage disorders
* Pregnant
* Any other laboratory abnormality, medical condition, or psychiatric disorders which in the opinion of the Investigator would put the subject's disease management at risk or may result in the subject being unable to comply with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-07-16 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Falone, MD, Study Director — American Regent, Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 41 study centers in the United States. The first subject was screened on 06 February 2014 and the last subject was completed on 07 July 2016.
Period: Overall Study
Arm/Group | Injectafer | Ferrous Sulfate Tablets
Started | 100 | 98
Completed | 92 | 85
Not Completed | 8 | 13
Not completed — Adverse Event | 1 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Study drug received outside protocol | 0 | 1
Not completed — Physician Decision | 4 | 0
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Population: Of the 198 subjects randomized, two subjects (one in each group) were not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Injectafer | Ferrous Sulfate Tablets | Total
Number analyzed (Participants) | 99 | 97 | 196
Age, Continuous [Median (Full Range); unit: years] | 38.3 [18.6 to 85.5] | 43.0 [18.5 to 74.3] | 40.5 [18.5 to 85.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 66 | 142
  Male | 23 | 31 | 54
Race/Ethnicity, Customized [Number; unit: participants] — Population: The category of Race is Check All That Apply. In the Injectafer group, two subjects didn't check any options and one subject checked two options. In the Oral Iron group, one subject checked two options.
  participants
    White: number analyzed (Participants) | 97 | 97 | 194
    White | 72 | 79 | 151
    Black/African American: number analyzed (Participants) | 97 | 97 | 194
    Black/African American | 25 | 17 | 42
    Asian: number analyzed (Participants) | 97 | 97 | 194
    Asian | 1 | 1 | 2
    American Indian/Alaska Native: number analyzed (Participants) | 97 | 97 | 194
    American Indian/Alaska Native | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 99 | 97 | 196
Point of Care Hemoglobin [Mean (Standard Deviation); unit: g/dL] — Population: Included subjects who received at least 1 dose of randomized treatment and had at least 1 post-randomization measurement of hemoglobin
  g/dL
    number analyzed (Participants) | 99 | 95 | 194
    (all) | 9.3 (1.19) | 9.4 (0.99) | 9.3 (1.10)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Screening Hepcidin and Change in Hemoglobin From Baseline to Highest Observed Hemoglobin Change (Proportion of Responders).
Description: Responders were defined as subjects achieving an increase from baseline ≥2 g/dL at anytime between baseline and the end of the study (Day 28). The relation between screening hepcidin and change in hemoglobin was assessed with regression models with baseline hepcidin and treatment group as independent factors. Treatment group differences (oral vs. IV iron) for mean changes in endpoints were assessed with the analysis of covariance with a fixed factor for treatment and baseline value as covariate. Treatment group differences for proportions were assessed with the normal approximation to the binomial distribution.
Time Frame: anytime between baseline and end of study (day 28) or time of intervention
Population: Full analysis set population
Measure: Count of Participants; unit: Participants
Arm/Group | Injectafer | Ferrous Sulfate Tablets
Number analyzed (Participants) | 94 | 92
Participants | 60 | 34

ADVERSE EVENTS:
Arm/Group | Injectafer | Ferrous Sulfate Tablets
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/97
Serious Adverse Events (participants affected / at risk) | 3/99 | 1/97
Other Adverse Events (participants affected / at risk) | 33/99 | 24/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectafer (N=99) | Ferrous Sulfate Tablets (N=97)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectafer (N=99) | Ferrous Sulfate Tablets (N=97)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Faeces discoulered (Gastrointestinal disorders) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Blood phosphorous decreased (Investigations) | 10 (10) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was stopped early due to slow enrollment, however it was not considered prematurely terminated. A total of 198 of the 400 subjects planned were randomized, 196 were treated, and the study concluded normally.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to publish the results collected from all sites. PI may publish results from a specific site if there is no multi-site publication within 12 months of the conclusion, abandonment or termination of the study. PI must provide sponsor with copy of draft publication at least 60 days before the scheduled submission to allow sponsor to protect confidential information. PI must withhold submission of publication for 90 days to allow sponsor to seek patent protection.